CLINICAL TRIAL: NCT02586038
Title: A MULTIARM, OPEN LABEL, RANDOMIZED PHASE II STUDY OF MLN9708 PLUS ORAL DEXAMETHASONE or PLUS ORAL CYCLOPHOSPHAMIDE AND DEXAMETHASONE or PLUS ORAL THALIDOMIDE AND DEXAMETHASONE FOLLOWED BY MAINTENANCE WITH MLN9708 IN NEWLY DIAGNOSED ELDERLY MULTIPLE MYELOMA PATIENTS
Brief Title: STUDY THAT COMPARE 3 ARM: MLN9708 DEXAMETHASONE, MLN9708 CYCLOPHOSPHAMIDE AND DEXAMETHASONE, MLN9708 THALIDOMIDE AND DEXAMETHASONE FOLLOWED BY MAINTENANCE WITH MLN9708 IN NEWLY DIAGNOSED ELDERLY MULTIPLE MYELOMA PATIENTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Boccadoro (Other)
Responsible Party: Sponsor-Investigator, Mario Boccadoro, Director, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNITO-EMN10
Record Dates: First submitted 2015-10-21; First posted 2015-10-26 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Dexamethasone; Cyclophosphamide; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MLN-DEX-CYCLO arm (Experimental): Patients will receive nine 28-days induction cycles.
  MLN9708: 4,0 mg orally on days 1, 8, 15 Dexamethasone: 40 mg orally on days 1, 8, 15, 22. Cyclophosphamide: 300 mg/sqm orally on days 1, 8, 15
  Interventions: Drug: MLN9708; Drug: Dexamethasone; Drug: Cyclophosphamide
- MLN-DEX-THAL arm (Experimental): Patients will receive nine 28-days induction cycles.
  MLN9708: 4,0 mg orally on days 1, 8, 15 Dexamethasone: 40 mg orally on days 1, 8, 15, 22. Thalidomide: 100 mg/day orally
  Interventions: Drug: MLN9708; Drug: Dexamethasone; Drug: Thalidomide

INTERVENTIONS:
Drug: MLN9708
Drug: Dexamethasone
Drug: Cyclophosphamide
  Arms: MLN-DEX-CYCLO arm
Drug: Thalidomide
  Arms: MLN-DEX-THAL arm

SUMMARY:
This study will evaluate the safety and the efficacy of the MLN-DEXAMETHASONE, MLN-DEXAMETHASONE-CYCLOPHOSPHAMIDE, or MLN- THALIDOMIDE-DEXAMETHASONE induction combinations, followed by MLN maintenance in newly diagnosed elderly Multiple Myeloma patients.

183 patients, males and females, older than 65 years old or younger but considered not eligible for high-dose chemotherapy and transplantation, enrolled in different sites, will take part in this study.

The duration of the study is approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal or surgically sterilized or willing to use two acceptable methods of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) for the duration of the study.
* Newly diagnosed MM based on standard CRAB criteria (see Appendix 12.2).
* Age ≥ 65 years old or younger not eligible for transplantation.
* Patient has measurable disease, defined as follows: any quantifiable serum monoclonal protein (M-protein) value (, ≥ 0.5 g/dL of M-protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours. For patients with oligo or non-secretory MM, it is required that they have measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan) or an abnormal free light chain ratio (n.v.: 0.26-1.65). We anticipate that less than 10% of patients admitted to this study will be oligo- or non-secretory MM with free light chains only in order to maximize interpretation of benefit results
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2
* Clinical laboratory values within 30 days of enrolment:

  * platelet count ≥ 75 x 109/L (Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment)
  * haemoglobin ≥ 8 g/dL
  * absolute neutrophil count (ANC) ≥ 1.0 x109/L
  * AST and ALT ≤ 3 times the upper limit of normal
  * total bilirubin ≤ 1.5 times the upper limit of normal
  * clearance creatinine ≥ 30 ml/min

Exclusion Criteria:

* Pregnant or lactating females.
* Serious medical condition, laboratory abnormality or psychiatric illness that prevented the subject from the enrolment or place the subject at unacceptable risk.
* Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid < to the equivalent of dexamethasone 40 mg/day for 4 days)
* Clinical active infectious hepatitis type A, B, C or HIV (HBV-DNA and HCV-RNA will be analysed to evaluate the cell proliferation of virus; anti-HIV antibody must be negative).
* Acute active infection requiring antibiotics or infiltrative pulmonary disease
* Peripheral neuropathy or neuropathic pain grade 2 or higher, as defined by National Cancer Institute Common Toxicity Criteria (NCI CTC) 4.03
* Contraindication to any of the required drugs or supportive treatments
* Invasive malignancy within the past 3 years
* Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort within 14 days before the first dose of study treatment (see Appendix 12.12).
* Diagnosis of Waldenstrom's macroglobulinemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2023-10 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Number of patients that will experience a progression disease after 2 years from diagnosis in 3 induction treatments, followed by maintenance with MLN9708, including:
  * MLN9708 plus dexamethasone (MLN-DEX)
  * MLN9708 plus dexamethasone and cyclophosphamide (MLN-CYCLO-DEX)
  * MLN9708 plus dexamethasone and thalidomide (MLN-THAL-DEX) A maximum of 61 patients per arm will be evaluated.

SECONDARY OUTCOMES:
Response rate | 5 years
  Response rate will evaluate efficacy in terms of Very Good Partial Remission (VGPR) of the 3 induction treatments, followed by maintenance with MLN9708. Rate of VGPR will be evaluated after cycle 4. Responses will be evaluated after each cycle.
  A maximum of 61 patients per arm will be evaluated.
Toxicity in terms of rate of hematologic and non-hematologic adverse events | 5 years
  Safety of combination will be evaluated in terms of rate of hematologic and non-hematologic adverse events of the 3 induction treatments, followed by maintenance with MLN9708. Toxicity will be evaluated according to the NCI CTCAE, version 4.03.
  A maximum of 61 patients per arm will be evaluated.
Progression Free Survival-2 (PFS-2) | 5 years
  Time from randomization to the date of first observation of second disease progression or death to any cause in each induction treatments A maximum of 61 patients per arm will be evaluated.
Time To Progression (TTP) | 5 years
  Time from the date of randomization to the date of first observation of progression, or deaths related to progression of the 3 induction treatments, followed by maintenance with MLN9708 A maximum of 61 patients per arm will be evaluated.
Time to Next Therapy (TNT) | 5 years
  Time from the date of randomization to the date of next anti-myeloma therapy of the 3 induction treatments, followed by maintenance with MLN9708 A maximum of 61 patients per arm will be evaluated.
Explorative comparative analyses | 5 years
  Explorative comparative analyses will be performed between the three arms and by in subgroups of patients, defined according to known prognostic factors A maximum of 61 patients per arm will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- AO SS Antonio e Biagio e Cesare Arrigo di Alessandria, Alessandria, Italy